CLINICAL TRIAL: NCT00878852
Title: Efficacy of a Contingency Management Program in the Treatment of Adolescents With Cannabis Use Disorders in a Child and Adolescent Psychiatry and Psychology Department
Brief Title: Efficacy of Contingency Management in the Treatment of Adolescents With Cannabis Use Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Javier Goti, Hospital Clinic Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI08/90331; 4363/2008 (Ethics Comitee HCP)
Record Dates: First submitted 2009-04-08; First posted 2009-04-09 (Estimated); Last update posted 2009-05-21 (Estimated); Status verified 2009-05

CONDITIONS: Marijuana Abuse
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard treatment (Active Comparator): Participants will be randomly assigned to a standard treatment group. Patients allocated to this group will receive active treatment in form of a 12-session intervention program. This program includes weekly intervention sessions developed according to the MET/CBT12 treatment protocol (Sampl, Kadden, 2001)
  Interventions: Behavioral: Standard treatment
- Experimental (Experimental): Participants randomly assigned to this group will received standard treatment (including 12 session therapy program) supplemented with an intervention with a contingency management program, designed to improve adherence and efficacy of the treatment program.
  Interventions: Behavioral: Standard Treatment Plus Contingency Management Program

INTERVENTIONS:
Behavioral: Standard treatment — Participants will be randomly assigned to a standard treatment group. Patients allocated to this group will receive active treatment in form of 12-session intervention program. This program includes weekly intervention sessions developed according to the MET/CBT12 treatment protocol (Sampl, Kadden, 2001). Intervention includes Motivational interviewing (2 sessions) and Cognitive behavioral therapy
  Arms: Standard treatment
Behavioral: Standard Treatment Plus Contingency Management Program — Participants assigned to this group will receive active treatment in form of 12-session intervention program. This program includes weekly intervention sessions developed according to the MET/CBT12 treatment protocol (Sampl, Kadden, 2001). Intervention includes Motivational interviewing (2 sessions) and Cognitive behavioral therapy (10 sessions). This treatment protocol will be supplemented with a contingency management intervention. Intervention will consist in a voucher program: negative urine-screens will be rewarded with vouchers. Voucher will have an increasing value. At the end of the program, vouchers can be changed by gifts. Potential gifts will be selected by the therapists and will be related to pro-social activities, aiming to change preexisting risk behaviours.
  Arms: Experimental

SUMMARY:
Cannabis use among Spanish adolescents has been increasing in the last decade. It has been related to poor school achievement, delinquency, substance use and psychiatric disorders. Furthermore, psychoactive substance use in adolescents presenting psychiatric disorders can result in the development of substance use disorders or the worsening of psychopathology. Thus, there's an urge to develop efficient interventions in the treatment of these disorders. Therapeutic approaches based on cognitive-behavioural therapy and motivational interviewing have demonstrated a limited efficacy in this population. Programs based on contingency management have been reported to be useful both in adult and adolescents, too. But it still remains unclear whether a combination of these therapeutic approaches is feasible and brings a better cost-benefit relation.

The investigators' project aims to evaluate the added benefits of supplementing a standard intervention on cannabis use, based on combined approach that includes motivational and cognitive-behavioural elements, with a contingency management program. Therefore, pre and post-treatment evaluation will be carried forward in a sample of 30 adolescents (aged 12-18) that initiate treatment for cannabis use related disorder at the Child and Adolescent Psychiatry Department of the Hospital Clinic in Barcelona. Participants will be randomly assigned to a standard treatment group or an experimental group in which standard treatment will be supplemented with a contingency management protocol. As a secondary objective, a prospective assessment of neuropsychological performance related to cannabis use or abstinence will be carried forward.

ELIGIBILITY:
Inclusion Criteria:

* Presence of DSM-IV-TR criteria of cannabis abuse and/or dependence
* Signed informed consent

Exclusion Criteria:

* Mental retardation
* Presence of a substance use disorder other than nicotine or cannabis
* Severe or unstable medical
* Presence at the moment of inclusion of severe acute psychopathology (acute psychotic symptoms, severe depressive symptoms, suicidal ideation)

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-04; Primary Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of marijuana active users | 12 weeks

SECONDARY OUTCOMES:
Percentage of negative urine-screens | 12 weeks
Percentage of completed intervention sessions | 12 weeks
Scores in psychopathology and drug scales (T-ASI, SDQ, BDI, Cannabis Problem Questionnaire) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Javier Goti, M.D, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic Barcelona, Barcelona, Barcelona, Spain

REFERENCES:
- [Background] Stephens RS, Babor TF, Kadden R, Miller M; Marijuana Treatment Project Research Group. The Marijuana Treatment Project: rationale, design and participant characteristics. Addiction. 2002 Dec;97 Suppl 1:109-24. doi: 10.1046/j.1360-0443.97.s01.6.x. PMID 12460133